CLINICAL TRIAL: NCT01669356
Title: The Effect of Parenteral Nutrition Supplement Versus Enteral Nutrition Alone on Nutrition Status After Esophagectomy: A Prospective Randomized Controlled Trial
Brief Title: The Effect of Parenteral Nutrition Supplement on Esophagectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNsupplESO; Energy Supply Trial (Other: Shanghai Zhongshan Hospital)
Record Dates: First submitted 2012-08-11; First posted 2012-08-21 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Esophagus Cancer
Keywords: malnutrition; parenteral supplement; rest metabolic rate; postoperative complications
MeSH Terms: conditions — Esophageal Neoplasms; Malnutrition; Postoperative Complications | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PN supplement (Experimental): Parenteral supplement with enteral nutrition for patients after esophagectomy
  Interventions: Other: Parenteral supplement with enteral nutrition for patients after esophagectomy
- EN alone (Active Comparator): Enteral nutrition alone for patients after esophagectomy
  Interventions: Other: Enteral Nutrition alone for patients after esophagectomy

INTERVENTIONS:
Other: Parenteral supplement with enteral nutrition for patients after esophagectomy
  Arms: PN supplement
Other: Enteral Nutrition alone for patients after esophagectomy
  Arms: EN alone

SUMMARY:
Malnutrition is common in esophagus cancer patients, especially after surgery therapy. Whether parenteral supplement with enteral nutrtion is benificial for patients after esophagectomy is controversial, when compared with enteral nutrition alone. In this study, the investigators are to examine the effect of enteral nutrition supplemented with parenteral nutrtion on nutrition status after esophagectomy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of esophagus cancer
* Undergo esophagectomy
* Nasoenteral tube is placed or surgical jejunostomy is performed

Exclusion Criteria:

* Contraindication for enteral nutrition or parenteral nutrition
* Malnutrition before surgery ( BMI > 30 or < 18.5)
* Hepatic dysfunction preoperatively
* Renal dysfunction preoperatively
* Infection before surgery
* Usage of corticosteroid before surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
postoperative laboratory parameters changes for nutrition assessment compared to preoperation | from one day before surgery to the 7th postoperative day
  plasma albumin, prealbumin, transferrin, retinaldehyde-binding protein, total lymphocytes counts
postoperative body composition change compared to preoperation measurement | from one day before surgery to the 7th postoperative day
  postoperative body composition is compared to preoperation, bioelectrical impedance spectroscopy is used for measurement of body composition

OTHER OUTCOMES:
complicatons incidence after surgery | 28 days after surgery
  complications involve anastomotic leakage, incision infection, pneumonia, catherter-related blood stream infection, respiratory failure

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, China

REFERENCES:
- [Derived] Wu W, Zhong M, Zhu DM, Song JQ, Huang JF, Wang Q, Tan LJ. Effect of Early Full-Calorie Nutrition Support Following Esophagectomy: A Randomized Controlled Trial. JPEN J Parenter Enteral Nutr. 2017 Sep;41(7):1146-1154. doi: 10.1177/0148607116651509. Epub 2016 May 20. PMID 27208039